CLINICAL TRIAL: NCT02665403
Title: Play Interventions to Reduce Anxiety and Negative Emotions in Hospitalized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KW/FR-12-020
Record Dates: First submitted 2016-01-17; First posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Play Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- play intervention (Experimental): 30 minutes of hospital play interventions
  Interventions: Other: Play intervention
- control (Placebo Comparator): usual care
  Interventions: Other: control

INTERVENTIONS:
Other: Play intervention — participants received around 30 minutes of hospital play interventions each day, conducted by hospital play specialists. Such interventions consisted of structured and non-structured activities. All these activities were given at the patients' bedside, with or without parental supervision, either once or spreading over an hour, depending on the ward routine.
  Arms: play intervention
Other: control — Children received standard medical and nursing care, such as vital signs observation, pharmacological treatment and wound and pain management as a control treatment
  Arms: control

SUMMARY:
Hospitalization is a stressful and threatening experience, which can be emotionally devastating to children. Hospital play interventions have been widely used to prepare children for invasive medical procedures and hospitalization. Nevertheless, there is an imperative need for rigorous empirical scrutiny of the effectiveness of hospital play interventions, in particular, using play activities to ease the psychological burden of hospitalized children. This study tested the effectiveness of play interventions to reduce anxiety and negative emotions in hospitalized children. A non-equivalent control group pre-test and post-test, between subjects design was conducted in the two largest acute-care public hospitals in Hong Kong. A total of 304 Chinese children (ages 3-12) admitted for treatments in these two hospitals were invited to participate in the study. Of the 304 paediatric patients, 154 received hospital play interventions and 150 received usual care.

DETAILED DESCRIPTION:
This study tested the effectiveness of play interventions to reduce anxiety and negative emotions in hospitalized children.

Intervention

Placebo control group

In the control group, children received standard medical and nursing care, such as vital signs observation, pharmacological treatment and wound and pain management.

Experimental group

In the experimental group, participants received around 30 minutes of hospital play interventions each day, conducted by hospital play specialists. The interventions in this study consisted of structured and non-structured activities. All these activities were given at the patients' bedside, with or without parental supervision, either once or spreading over an hour, depending on the ward routine.

Data Collection Methods

Approval for the study was obtained from the hospital ethics committees. A research assistant collected demographic data from the parents and from the children's medical records after obtaining the consent form. The children's baseline anxiety levels were also documented. For the experimental group, the interventions started after the baseline data had been collected. The emotional behaviour of each child was observed by a research assistant for two consecutive days, at the end of which a research assistant documented the child's overall emotional behaviour, using the CEMS. The child's anxiety levels were reassessed and documented.

Analysis

The Statistical Package for Social Science (SPSS) software, version 20.0 for Windows was used for the data analysis. Descriptive statistics were used to calculate the means, standard deviations, and ranges of the scores on the various scales. The homogeneity of the two groups was examined using inferential statistics (independent t-test and chi-squared). The interrelationships among the scores on the different scales and the demographic variables were assessed using the Pearson product-moment correlation coefficient. Differences in the mean scores on the CEMS and the children's anxiety levels between the two intervention groups were investigated by an independent t-test and mixed between-within subjects ANOVA, respectively. Multiple regression analysis was performed to examine the effects of participants' demographic and clinical characteristics on the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* were Chinese children aged between 3 and 12,
* able to speak Cantonese
* required to stay in hospital for at least three consecutive days

Exclusion Criteria:

* children with identified cognitive and learning difficulties

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Anxiety levels change from baseline at 2 days after admission between intervention and control group for children aged 3 - 7 | two days after admission
  Anxiety levels of children aged between 3 and 7 were assessed by using the Visual Analogue Scale , which consists of a 10 cm horizontal line on a piece of card, with different facial expressions supplemented by the words 'I have no anxiety' at one end and 'I have so much anxiety' at the other. They were asked to respond to this scale at 2 days after admission.

SECONDARY OUTCOMES:
Anxiety levels change from baseline at 2 days after admission between intervention and control group for children aged 8 - 12 | two days after admission
  Anxiety levels of children aged between 8 and 12 were assessed by using the short-form Chinese version of the State Anxiety Scale for Children (CSAS-C). This consists of 10 items scored from 1 to 3, with total scores ranging from 10 to 30. Higher scores represent greater anxiety. They were asked to respond to this scale at 2 days after admission.
baseline anxiety levels for children aged 3 - 7 | baseline
  Anxiety levels of children aged between 3 and 7 were assessed by using the Visual Analogue Scale , which consists of a 10 cm horizontal line on a piece of card, with different facial expressions supplemented by the words 'I have no anxiety' at one end and 'I have so much anxiety' at the other. They were asked to respond to this scale at baseline .
baseline anxiety levels for children aged 8 -12 | baseline
  Anxiety levels of children aged between 8 and 12 were assessed by using the short-form Chinese version of the State Anxiety Scale for Children (CSAS-C). This consists of 10 items scored from 1 to 3, with total scores ranging from 10 to 30. Higher scores represent greater anxiety. They were asked to respond to this scale at baseline.
overall emotion behaviors for the 2-day period of hospitalization (CEMS) | the 2-day period of hospitalization
  The emotions of the hospitalized children were assessed using the Children's Emotional Manifestation Scale (CEMS), which is an observation scale. The CEMS consists of five categories, each category scored from 1 to 5, with summed scores from 5 to 25. Higher scores represent more negative emotional behavior. The emotional behaviour of each child was observed by a research assistant for two consecutive days, at the end of which a research assistant documented the child's overall emotional behaviour, using the CEMS.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung, William LI, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan for making the data available to the public

REFERENCES:
- [Derived] Li WHC, Chung JOK, Ho KY, Kwok BMC. Play interventions to reduce anxiety and negative emotions in hospitalized children. BMC Pediatr. 2016 Mar 11;16:36. doi: 10.1186/s12887-016-0570-5. PMID 26969158